CLINICAL TRIAL: NCT05979766
Title: Effects of Manual Lymphatic Drainage Versus Marian Clark Drainage on Pain and Disability in Patients With Pelvic Congestion Syndrome
Brief Title: Manual Lymphatic Drainage vs Marian Clark Drainage in Pcs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIUmib
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Congestive Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual lymphatic drainage vs marian clark drainage (Active Comparator): Effect of Marian Clark drainage and manual lymphatic drainage in women suffering from pelvic congestion syndrome
  Interventions: Other: Manual lymphatic drainage versus marian clark drainage
- Manual lymphatic drainage versus marian clark drainage (Active Comparator): Effect of Marian Clark drainage and manual lymphatic drainage in women suffering from pelvic congestion syndrome
  Interventions: Other: Manual lymphatic drainage versus marian clark drainage

INTERVENTIONS:
Other: Manual lymphatic drainage versus marian clark drainage — Manual lymphatic drainage versus marian clark drainage

SUMMARY:
Pelvic congestion syndrome is a debilitating and potentially life threatening disorder of the pelvic region there is a constant hindrance in patient's daily professional and personal life due to the chronic pain. it can provide a definite way to improve pelvic congestion and quality of life. In this way it can benefit a large percentage of community females suffering from pelvic congestion syndrome and disability. This can grow at large length in favour of patients, clinicians and overall women health.

DETAILED DESCRIPTION:
As per researcher's knowledge there are limited researches in which efficacy of manual lymphatic drainage in pelvic congestion syndrome are analyzed furthermore my comparative intervention i.e Marian Clark drainage is a rarely used osteopathic technique and not much studies have been conducted on it. This study helped to in identifying the effect of manual lymphatic drainage versus Marian Clark drainage on pain and disability in patients with pelvic congestion syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous women
* Age ranging 20 to 50
* Ovarian veins >4mm in diameter on Ultrasound Chronic pelvic pain/pressure for more than 6 months.
* Dull, aching or "dragging" pain in the pelvis or lower back, particularly on standing and worse around the time of your menstrual period.
* Pelvic pain that worsens as the day goes on, particularly if much time is spent standing dyspareunia
* Swollen veins in pelvic region, butt, thighs, vulva and vagina.
* Associated Irritable bladder/Irritable bowel present

Exclusion Criteria:

* Pelvic pain due to other organic cause like uterine fibroids, Endometriosis, Ovarian cyst pelvic pain due to neurological or musculoskeletal disorder
* Uterine prolapse
* Pelvic cancer

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Manual lymphatic drainage | 6 months
  Treatment protocol to group A
  It consists of 15 patients who will receive manual lymphatic drainage 4 sessions per week for 12 weeks
  Manual Lymph Drainage Techniques for Pelvic Decongestion
  Step 1: short neck treatment (supraclavicular fossa or SCF)
  Step 2: (two parts: visceral, deep)
  Visceral:
  Deep: Treatment of the thoracic duct, cisterna Chyli
  Deep Abdominal Manual lymphatic drainage
  Step-3. Treatment of right Axillary Lymph nodes
  Step-4. Establish the Right inguino-Axillary Anastomosis.
  Step-5. Decongest the right ipsilateral lower abdomen and suprapubic area
  Step-6 Treatment of Left Axillary Lymph nodes
  Step-7. Establish the Left inguino-Axillary Anastomosis.
  Step-8. Decongest the Let ipsilateral lower abdomen and suprapubic area
Marian clark drainage | 6 months
  It consists of 15 patients who will receive Marian clark drainage 4 sessions per week for 12 weeks each session will continue till therapist feels palpable change in congestion in pelvic area medial to Anterior superior Iliac spine.
  * Stand to the side of the patient
  * Patient semiprone on all fours
  * Hook fingers medial to both Anterior superior Iliac spine
  * Pull hands cephalad (traction)
  * Patient arches back like a cat
  * Encourage this movement with cephalad rocking
  * Repeat for several minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam Muneeb, Ms, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No